CLINICAL TRIAL: NCT01491282
Title: Brown Adipose Tissue After Vagus Nerve Stimulation
Brief Title: Study of the Effect of Vagus Nerve Stimulation on Human Brown Adipose Tissue Activity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University (Other)
Responsible Party: Principal Investigator, dr. Sef Janssen, Dr. W.D. van Marken Lichtenbelt, Maastricht University
Other Study IDs: MEC 10-3-071
Record Dates: First submitted 2010-11-30; First posted 2011-12-13 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Obesity
Keywords: human brown adipose tissue activity; obesity; energy metabolism; adaptive thermogenesis
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment
  Interventions: Other: Enabling and disabling VNS

INTERVENTIONS:
Other: Enabling and disabling VNS — No intervention
  Other Names: VNS

SUMMARY:
To evaluate the effect of vagus nerve stimulation for refractory epilepsy on the activity of human brown adipose tissue.

ELIGIBILITY:
Inclusion Criteria:

* Subjects treated with VNS for epilepsy, aged 18-65 years, with a Body Mass Index (BMI) ≤ 28 kg/m2.

Exclusion Criteria:

* Body Mass Index > 28 kg/m2
* Daily epileptic insults.
* Subjects that need 'Rapid Cycling' VNS to control their frequency of epileptic insults.
* Psychological unstable subjects (as judged by the treating neurologist).
* subjects with mental retardation (as judged by the treating neurologist).
* subjects with severe behaviour disorders (as judged by the treating neurologist).
* Pregnant subjects.
* Subjects that previously underwent high dose radiation for diagnostic or therapeutic purposes (radiotherapy, high frequency CT-scans).
* The use of the following medication is an exclusion criterium;

  * ß-blockers,
  * Ketogenic diet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postoperative patients treated with vagus nerve stimulation for refractory epilepsy
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
human brown adipose tissue activity | baseline and 2 weeks after

CONTACTS AND LOCATIONS:
Overall Officials: Wouter D. van Marken Lichtenbelt, PhD., Principal Investigator — Department of Human Biology, Maastricht University
Locations (1):
- Maastricht University, Maastricht, Netherlands

REFERENCES:
- [Derived] Vijgen GH, Bouvy ND, Leenen L, Rijkers K, Cornips E, Majoie M, Brans B, van Marken Lichtenbelt WD. Vagus nerve stimulation increases energy expenditure: relation to brown adipose tissue activity. PLoS One. 2013 Oct 23;8(10):e77221. doi: 10.1371/journal.pone.0077221. eCollection 2013. PMID 24194874